CLINICAL TRIAL: NCT05631587
Title: A Technology-based Intervention for Promoting Physical Activity Among Post-treatment Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: University of Victoria (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 21485
Record Dates: First submitted 2022-11-07; First posted 2022-11-30 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Survivorship
Keywords: cancer survivor; physical activity; website
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: A two-arm, assessor-blinded RCT examining the effect of a website for physical activity promotion in cancer survivors (WExercise)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (WExercise) (Experimental): Participants will receive a written information sheet (i.e., PA guide, safety precautions, and goal) same as the control group. In addition, participants in the WExercise group will be provided with 10 weekly technology-based classes delivered in a mobile application aimed at promoting PA. Participants will be given individualised access to the app. The classes aim at developing reflective, regulatory, and reflexive processes of cancer survivors to engage in PA based on the M-PAC framework. Participants will be sent reminders (3 days apart) by WhatsApp/WeChat each time they have a class due.
  Interventions: Behavioral: WExercise
- Control condition (Self-directed exercise) (Active Comparator): Participants will receive a one-page written information sheet regarding the PA guidelines for cancer survivors and exercise safety precautions extracted from the website of the Centre for Health Protection of the HKSAR Government. Although mixed aerobic and resistance exercise are recommended, participants will be provided with a simple goal of increasing their aerobic exercise levels to 150 minutes of moderate aerobic activity or 75 minutes of vigorous aerobic exercise per week because resistance exercise requires instructions from trained personnel.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: WExercise — A 10-weekly technology-based intervention delivered in a mobile application using the M-PAC framework to promote PA in post-treatment cancer survivors. Participants will be given individualised access to the app. Participants will be sent reminders (3 days apart) by WhatsApp/WeChat each time they have a class due.
  Arms: Intervention condition (WExercise)
Behavioral: Control — A control group receiving an information sheet for self-directed exercise.
  Arms: Control condition (Self-directed exercise)

SUMMARY:
Cancer survivors generally have low physical activity (PA) levels. While literature shows some evidence of improvement in PA following technology-based PA promotion interventions among cancer survivors, high-quality randomised control trials (RCTs), with objective measures of PA and longer-term follow-up, are lacking. Using a theoretical framework that addresses action control in addition to intention formation may enhance intervention effect. The Multi-process action control (M-PAC) framework is an extension of the traditional intention-formation theories, incorporating constructs that address the translation of intention into behaviour and continual action control. After comprehensively searching, no previous or ongoing RCTs have investigated the efficacy of a technology-based PA promotion intervention in cancer survivors that is designed based on the M-PAC framework. Investigators therefore propose a RCT to evaluate a technology-based intervention (WExercise) to support the promotion of PA in cancer survivors.

DETAILED DESCRIPTION:
Objective: To develop a technology-based physical activity promotion intervention (WExercise) for cancer survivors based on the Multi-process Action Control (M-PAC) Framework and examine its usability and efficacy.

Main hypothesis: The WExercise group will have a significantly greater increase in aerobic exercise than the self-directed exercise group at post-intervention.

Design: Phase 1- Application development; Phase 2- Usability testing (n=10); Phase 3- Assessor-blind two-arm randomized controlled trial (n=98; WExercise or self-directed exercise group).

Subjects: Physically inactive cancer survivors who have completed curative treatment.

Study instruments: Accelerometry, Godin Leisure Time Exercise Questionnaire, 6-minute walk test, EORTC QLQ-C30, M-PAC questionniare; administered at baseline, post-intervention, and 3 months post-intervention.

Interventions: Both groups will receive written physical activity guidelines with a goal to engage in at least 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity aerobic exercise per week. The WExercise group will additionally receive 10 weekly automated online classes delivered on a mobile application which aim at developing participants' reflective, regulatory, and reflexive processes based on the M-PAC to achieve recommended physical activity levels (1st-3rd week: intention formation; 4th-8th weeks: behavioral regulations; 9th-10th weeks: action control maintenance).

Main outcomes: Time spent in moderate-to-vigorous aerobic exercise (primary), exercise capacity, and quality of life.

Data analysis: Intention-to-treat analysis will be performed. Application usage in the WExercise group will be presented in descriptive statistics. Generalized linear mixed-effect models will be used to assess between-group and within-group differences in the outcomes.

Expected results: The findings will inform the design of future eHealth interventions to encourage and sustain health behavior change in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* completion of primary treatment (surgery/chemo-/radiation therapy) of curative intent for at least 12 months,
* no metastasis, no recurrence
* not meeting the recommended PA guideline (<150 min of moderate intensity aerobic exercise and <75 min of vigorous aerobic exercise per week)
* access to Internet
* able to read Chinese and communicate in Cantonese or Putonghua
* screened by a nurse as no contraindications for engaging in unsupervised exercise using a risk screening tool

Exclusion Criteria:

* have a psychiatric disorder
* significant cognitive impairment
* a history of more than one cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in aerobic exercise behaviour (objective measure) | Measure at Baseline (Week 0), Post-intervention (Week 11), 3 months post-intervention (Week 23). Each time point will measure 7 full consecutive days and average time (minutes) per day spent in moderate-to-vigorous aerobic exercise will be reported.
  Measured as time spent in moderate-to-vigorous aerobic exercise using accelerometer
Change in aerobic exercise behaviour (subjective measure) | Measure at Baseline (Week 0), Post-intervention (Week 11), 3 months post-intervention (Week 23). Self-reported minutes of moderate-to-vigorous aerobic exercise will be recorded.
  Measured by the Godin Leisure Time Exercise Questionnaire (Min and Max NA; higher scores represent higher aerobic exercise level)

SECONDARY OUTCOMES:
Change in exercise capacity | Measure at Baseline (Week 0), Post-intervention (Week 11), 3 months post-intervention (Week 23).
  Measured by the 6-minute walk test to estimate the peak oxygen uptake
Change in cancer-specific Quality of life | Measure at Baseline (Week 0), Post-intervention (Week 11), 3 months post-intervention (Week 23).
  Measured by the 30-item European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) to estimate the general well-being of cancer patients. The score ranges from 0-100, a high score for a functional scale represents a healthy level of functioning; a high score for the global health status / QoL represents a high QoL; but a high score for a symptom scale / item represents more severe symptoms.
Change in key components of M-PAC framework | Measure at Baseline (Week 0), Mid-intervention (Week 5), Post-intervention (Week 11), 3 months post-intervention (Week 23).
  Measured by the Multi-Process Action Control (M-PAC) questionnaire. The following components will be measured in 5-point Likert scale: affective attitude (score:3-15), instrumental attitude(score:3-15), perceived capability (score:3-15), perceived opportunity (score:3-15), behavioural regulation (score:6-30), habit formation (score:4-20), identity formation (score:4-20); and two items for decisional intentions (score:1-12). Higher score means higher levels of reflective, regulatory, and reflexive processes that may have facilitated exercise behavior change.
Application usage | Measure at post-intervention (Week 11)
  Reported as the number of interventional classes completed using inbuilt tracking tools.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes RE. Chapter Five - The Evolving Understanding of Physical Activity Behavior: A Multi-Process Action Control Approach. In: Elliot AJ, editor. Advances in Motivation Science. 4: Elsevier; 2017. p. 171-205.
- [Background] Gutteridge JM, Toeg D. Iron-dependent free radical damage to DNA and deoxyribose. Separation of TBA-reactive intermediates. Int J Biochem. 1982;14(10):891-3. doi: 10.1016/0020-711x(82)90071-4. PMID 6290280